CLINICAL TRIAL: NCT03828929
Title: Effect of IV Vitamin C, Thiamine, and Steroids on Mortality of Septic Shock
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recent similar studies have been completed and published showing no benefit to the intervention.
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Responsible Party: Principal Investigator, Liam Gross, Instructor of Clinical Medicine, Principle Investigator, New York Presbyterian Brooklyn Methodist Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1220432
Record Dates: First submitted 2019-01-29; First posted 2019-02-04 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Ascorbic Acid; Thiamine; Saline Solution; Glucose

STUDY DESIGN:
Intervention Model Description: Study is performed with 2 arms, interventional arm with thiamine and vitamin C, and the control arm with placebo in a 1:1 ratio.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pharmacist who prepares the medication is in charge of blinding randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vitamin C and Thiamine (Experimental): IV vitamin C, 1500mg in 50ml of normal saline every six hours, infused over one hour and IV Thiamine 200mg in 50ml of 5% dextrose every 12 hours, for 4 days or until discharge from the intensive care unit, whichever comes first.
  Interventions: Drug: Vitamin C
- Placebo (Placebo Comparator): 50ml of IV normal saline every six hours and 50ml of IV 5% dextrose every 12 hours, for 4 days or until discharge from the intensive care unit, whichever comes first.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Vitamin C — IV vitamin C, 1500mg in 50ml of normal saline every six hours, infused over one hour and IV Thiamine 200mg in 50ml of 5% dextrose every 12 hours, for 4 days or until discharge from the intensive care unit, whichever comes first.
  Other Names: Thiamine
  Arms: Vitamin C and Thiamine
Drug: Normal saline — 50ml of IV normal saline every six hours and 50ml of IV 5% dextrose every 12 hours, for 4 days or until discharge from the intensive care unit, whichever comes first.
  Other Names: 5% dextrose
  Arms: Placebo

SUMMARY:
Preliminary studies show that giving a "cocktail" of intravenous vitamin C, vitamin B1, and steroids to critically ill patients with septic shock may dramatically improve mortality in those patients. These studies suffer from inadequate design due to lack of controls and blinding to prove the causal effect. Our goal is to conduct a prospective blinded randomized control trial to investigate whether this intervention truly effect outcomes.

DETAILED DESCRIPTION:
This is a double-blind randomized placebo controlled study. Only the dispensing pharmacist, who has no clinical interaction with the patient and is not part of the bedside treatment team, will be aware of the treatment allocation. Patients will be randomized into one of 2 groups: the intervention group and the control group. Intervention group will receive intravenous vitamin C and thiamine according to the dosing regimen described below. The control group will receive placebo that is prepared to look identical to the medications within the intervention group.

Randomization will be performed using a random number table generated by the dispensing pharmacist using randomization software. The software will generate subject Identification numbers (IDs) from 1 to 130 and randomize half of the IDs to the control and half to the treatment group. The table will be generated prior to enrollment of the first participant. Once enrollment begins, each participant's medical record number (MRN) will be assigned to the subject IDs in sequential order from 1 to 130. This process will be triggered by the fellow ordering the vitamin C protocol. Only the pharmacist will have access to the table(which will be stored securely) until completion of the study.

The hydrocortisone, vitamin C, thiamine, and their corresponding placebos will be formulated as follows:

Vitamin C: Vitamin C is provided by the manufacturer as a 50ml vial at a concentration of 500mg/ml. Three (3) ml of vitamin C will be placed in a 50 ml bag of Normal Saline (1500mg vitamin C in 50ml bag) which will then be infused over 1 hour. The bag will be labeled by the pharmacy as Vitamin C. The dosing schedule is 1500mg every 6 hours for 4 days or until discharge from the ICU.

Vitamin C placebo will consist of an identical bag of 50cc normal saline (but with no vitamin C) and will be labelled vitamin C. Placebo will be infused over 30-60 minutes as per the infusion instructions of the active vitamin.

Thiamine: As a high percentage of septic patients have been shown to be thiamine deficient, patients will receive intravenous thiamine 200mg q 12 hourly for 4 days or until ICU discharge. Thiamine is also a cofactor for the metabolism of oxalate (a byproduct of vitamin C metabolism), with thiamine deficiency increasing oxalate levels. Thiamine placebo will consist of 50mL of 5% dextrose.

Steroids: Hydrocortisone 50 mg IV q 6 hourly will be continued for at least 4 days or until ICU discharge. All patients(both in the treatment and the control groups) included in the study will receive this steroid regimen. If participants were already started on steroids for another indication (i.e Asthma) prior to inclusion, they may continue their regimen as long as the dosing is equivalent to the steroid regimen described above. Alternatively, dosing may need to be increased or regimen switched entirely to the one described in this protocol. This decision will be made by the treating physician.

Procalcitonin will be drawn at time of admission and again at 96 hours after admission.

Patients who are enrolled in the study will have their capillary blood glucose levels measured using the StatStrip Glucometer and Test Strips. This glucometer is currently being used for all patients at NYPBMH.

Data collection: data collection will be performed by the research associate and other study personnel in real time and as the schedule allows. The data collection sheet (see Appendix) will include all needed data associated with the patient's MRN. Once the data sheet is completed, the patient's treatment group can be unmasked - this will occur after the 60 day mark, as that is the last data point (60-day mortality).

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to medical intensive care unit (MICU) for less than 24 hours, who are hypotensive despite a fluid bolus of 30 mL/kg and who are requiring pressors to keep MAP > 65 of at least 5 mcg/min of levophed or equivalent and whose shock is clinically suspected to be secondary to sepsis.
* In addition, stress dose corticosteroids, hydrocortisone 50mg IV Q6hrs, will have to have been started or intended to be started.

Exclusion Criteria:

* Contraindication to corticosteroids, thiamine, or vitamin C
* Treating physician opposed to administering corticosteroids to the patient
* Age < 18 years
* Pregnancy
* DNR/DNI/limitations of care
* Patients with a fatal underlying disease who are unlikely to survive to hospital discharge
* Patients with a primary admitting diagnosis of an acute cerebral vascular event, acute coronary syndrome, active gastrointestinal bleeding, burn or trauma
* Requirement for immediate surgery
* Patients with HIV and a CD4 < 50 mm2
* Patients with known glucose-6 phosphate dehydrogenase (G-6PD) deficiency.8
* Involvement in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-01-28 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Hospital Mortality | All Cause in Hospital Mortality average 30 days
  In Hospital Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Liam Gross, DO, Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Marik PE, Khangoora V, Rivera R, Hooper MH, Catravas J. Hydrocortisone, Vitamin C, and Thiamine for the Treatment of Severe Sepsis and Septic Shock: A Retrospective Before-After Study. Chest. 2017 Jun;151(6):1229-1238. doi: 10.1016/j.chest.2016.11.036. Epub 2016 Dec 6. PMID 27940189

DOCUMENTS (1):
  • Study Protocol (2019-01-15): https://cdn.clinicaltrials.gov/large-docs/29/NCT03828929/Prot_000.pdf